CLINICAL TRIAL: NCT01707225
Title: Safety and Efficacy of Octreotide LAR Depot in Left Ventricular Assist Device (LVAD) Associate Gastrointestinal (GI)
Brief Title: Safety Study of Octreotide Injection to Prevent GI Bleeding in Patients With Left Ventricular Assist Device (LVAD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Thoratec Corporation (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM14516
Record Dates: First submitted 2012-10-11; First posted 2012-10-16 (Estimated); Results first posted 2016-01-12 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2016-12

CONDITIONS: Gastrointestinal Bleeding
Keywords: GI Bleeding; Gastrointestinal bleeding; LVAD
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Octreotide LAR Depot (Experimental): Once enrolled in the study subjects will receive a monthly intra-muscular injection of 20mg of octreotide LAR at each study visit for 24 weeks and will be followed for a total of 36 weeks.
  Interventions: Drug: Octreotide LAR Depot

INTERVENTIONS:
Drug: Octreotide LAR Depot — The subject will be seen in clinic every 4 weeks (+/- 4 days) through week 24. During weeks 25-36 the subject will receive a telephone call every 4 weeks +/- 4 days, from the research nurse to assess for changes occurring after the study drug was stopped. Subjects will receive a physical exam and interview at each visit to assess for any sign of GI bleeding at home as per standard protocol for HeartMate II patients and for potential drug related side effects. Labs collected for research will include monthly basic metabolic panel (BMP), complete blood count (CBC), fructosamine and quarterly HGbA1C , VEGF, vWF, vWF activity assay, thyroid stimulating hormone (TSH), platelet function test and fibrinogen. Subjects will receive their monthly injection while in clinic for their every 4 weeks appointment. The subjects will be followed and data will be collected for 36 weeks, or for as long as they are enrolled in the study.

SUMMARY:
The investigators hypothesize that octreotide LAR (Long Acting Release) safely decreases GI bleeding in patients with a left ventricular assist device (LVAD). Patients undergoing implantation of non-pulsatile, continuous-flow LVAD have a higher incidence of gastrointestinal bleeding. This is a significantly associated morbidity and can threaten a patient's life as well as their ability to undergo eventual heart transplantation secondary to both general health/strength and the potential development of antibodies to blood products that would make future transfusions and transplantations more difficult.

If this research finds that use of octreotide LAR can decrease the incidence of gastrointestinal bleeding in this patient population, it will revolutionize the manner in which these patients are managed. The finding of reduced GI bleeding would allow the patient to have less exposure to blood products, reduce hospitalizations, and ensure that subsequent transplant planning not be delayed. This would not only be of great benefit to the patient, but would significantly decrease health-care costs through preventive measures.

The goal of this project is to study whether the regular administration of monthly octreotide LAR is safe and if it will decrease the incidence of gastrointestinal bleeding in patients undergoing implantation of non-pulsatile, continuous flow left ventricular assist devices (LVAD).

DETAILED DESCRIPTION:
The primary specific aim is to determine the safety of octreotide LAR in patients with a LVAD.

Patient experience of the following will be assessed throughout the study (list obtained from up-to-date.com)

Cardiovascular:

Sinus bradycardia (19% to 25%) Hypertension (≤13%) conduction abnormalities (9% to 10%)

Central nervous system:

Fatigue (1% to 32%) headache (6% to 30%) malaise (16% to 20%) fever (16% to 20%) dizziness (5% to 20%) Pain (4% to 15%)

Dermatologic:

Pruritus (≤18%) Rash (15%; depot formulation) alopecia (≤13%)

Endocrine & metabolic:

Hyperglycemia (2% to 27%)

Gastrointestinal:

Abdominal pain (5% to 61%) loose stools (5% to 61%) nausea (5% to 61%) diarrhea (34% to 58%) flatulence (≤38%) cholelithiasis (13% to 38%; length of therapy dependent) constipation (9% to 21%) vomiting (4% to 21%)

Hematologic Anemia (5-15%)

Local:

Injection site pain (2% to 50%; dose and formulation related)

Neuromuscular & skeletal:

Back pain (1% to 27%) arthropathy (8% to 19%) myalgia (≤18%)

Renal Kidney Stones (5-15%)

Respiratory:

Upper respiratory infection (10% to 23%)

Miscellaneous:

flu symptoms (1% to 20%)

Our key secondary outcomes will focus on study drug efficacy. Patient experience of the following will be assessed:

Need for Blood Transfusion Hospital Admission for GI Bleed

Heart disease is a leading cause of death and disability, according to the American Heart Association. Current therapies include lifestyle modification, medical management and revascularization via Percutaneous Coronary Intervention (PCI) or Coronary Artery Bypass Surgery (CABG). However, a large portion of patients develop cardiomyopathy which is refractory to the above interventions. They are treated with chronic inotropes, resynchronization and other forms of medical management.

Many of these patients eventually worsen and need consideration for cardiac transplantation. The Thoratec Heartmate II, which is the primary left ventricular assist device (LVAD) implanted at our institution, has been used as a bridge-to-transplantation. More recently it has been approved as destination therapy for patients who are not candidates for transplantation. Over 6000 of these devices have been implanted worldwide since their introduction. We have implanted over 70 here at the VCU Health System and the McGuire VA Medical Center.

The early LVAD devices provided physiologic pulsatility, but were large in size and required large catheters for external venting. The newer continuous flow LVAD devices, such as the Heartmate II, offer the benefit of being smaller and easier to implant as well as improving mobility and thus quality of life. However, this benefit comes with a complication of an increased incidence of GI bleeding, thought to be related to the loss of pulsatility and the nature of these smaller devices.

Approximately 10-30% of patients experience at least one episode GI bleeding which is likely multifactorial. It has already been demonstrated that an acquired von Willebrand Syndrome (vWS) develops due to destruction of multimeric vWF. Additionally, it has been shown that these patients have a higher than normal percentage of gastrointestinal angiodysplasia. Whether these are preexisting or develop as a result of de novo angiogenesis from the gut mucosa is unknown. It is thought that the loss of pulsatility and potential hypoxia result in secretion of angiogenic mediators and contribute to the development of angiodysplasia.

Current treatment for LVAD associated GI bleeding is aimed at identifying the location of bleeding and treatment with blood product transfusion, cryoprecipitate for vWS, Desmopressin for platelet dysfunction, and interventions through Interventional Radiology (IR) and surgery. In addition to the obvious costs and increase in morbidity and mortality associated with the above therapies, patients who receive multiple transfusions develop antibodies and thus become more difficult to transplant. Thus a vicious cycle develops.

We need to strive for a proactive stance in these patients and attack the problem at the source. There is a considerable amount of experience using octreotide in idiopathic chronic GI bleeding. This is likely due to its ability to decrease splanchnic blood flow and its potential ability to inhibit angiogenesis. Octreotide has been thoroughly studied and has a known safety profile. Off label use of octreotide LAR for the purpose of attenuating LVAD associated GI bleeding is currently practiced by some physicians at VCU with no adverse side effects encountered. It is time to formally study the safety and efficacy of octreotide LAR for this purpose. We propose an open-label safety study for 10 subjects to be followed for a total of 24 weeks. Should the safety study be favorably completed, a multi-center trial with randomization to octreotide LAR or placebo with endpoints of GI bleeding and transfusion will be pursued.

ELIGIBILITY:
Inclusion Criteria:

* LVAD insertion as bridge to transplant or destination
* 18 years of age or older

Exclusion Criteria:

* Poorly controlled diabetes, A1C greater than 8%
* Poorly controlled hypothyroidism, TSH > upper limit of normal (5.5)
* End Stage Renal Disease (ESRD) requiring dialysis
* Cirrhosis
* Anemia (Hgb < 8)
* Acromegaly
* Hx of chronic diarrhea - as determined by history of loose stool lasting longer than 2-4 weeks
* Pregnancy or breastfeeding
* Inability to provide informed consent
* Incarceration or otherwise a ward of the state
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Malhotra, DO MS, Principal Investigator — VCU
Locations (1):
- Virginia Commonwealth University Health System, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Octreotide LAR Depot: Once enrolled in the study subjects will receive a monthly IM injection of 20mg of octreotide LAR at each study visit for 24 weeks and will be followed for a total of 36 weeks.
  Octreotide LAR Depot: subject seen in clinic every 4 weeks (+/- 4 days) through week 24. Weeks 25-36 subject will receive a call every 4 weeks +/- 4 days, to assess for changes after the study drug was stopped. Subjects will receive a exam and interview at each visit to assess for GI bleeding at home and for drug related side effects. Labs collected for research will include monthly basic metabolic panel (BMP), complete blood count (CBC), fructosamine and quarterly HGbA1C , VEGF, vWF, vWF activity assay, thyroid stimulating hormone (TSH), platelet function test and fibrinogen. Subjects will receive their monthly injection while in clinic for their every 4 weeks appointment. The subjects will be followed and data will be collected for 36 weeks, or for as long as they are enrolled in the study.
Period: Overall Study
Arm/Group | Octreotide LAR Depot
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Octreotide LAR Depot
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 2
Gender [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Side-Effects
Description: Cardiovascular:
  Sinus bradycardia (19% to 25%) Hypertension (≤13%) conduction abnormalities (9% to 10%)
  Central nervous system:
  Fatigue (1% to 32%) headache (6% to 30%) malaise (16% to 20%) fever (16% to 20%) dizziness (5% to 20%) Pain (4% to 15%)
  Dermatologic:
  Pruritus (≤18%) Rash (15%; depot formulation) alopecia (≤13%)
  Endocrine & metabolic:
  Hyperglycemia (2% to 27%)
  Gastrointestinal:
  Abdominal pain (5% to 61%) loose stools (5% to 61%) nausea (5% to 61%) diarrhea (34% to 58%) flatulence (≤38%) cholelithiasis (13% to 38%; length of therapy dependent) constipation (9% to 21%) vomiting (4% to 21%)
  Hematologic Anemia (5-15%)
  Local:
  Injection site pain (2% to 50%; dose and formulation related)
  Neuromuscular & skeletal:
  Back pain (1% to 27%) arthropathy (8% to 19%) myalgia (≤18%)
  Renal Kidney Stones (5-15%)
  Respiratory:
  Upper respiratory infection (10% to 23%)
  Miscellaneous:
  flu symptoms (1% to 20%)
Time Frame: 24 weeks
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Octreotide LAR Depot
Number analyzed (Participants) | 10
participants | 10 [0 to 10]

2. Secondary Outcome: Need for Blood Transfusion and Hospital Admission for GI Bleed
Time Frame: 24 weeks
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Octreotide LAR Depot
Number analyzed (Participants) | 10
participants | 10 [0 to 10]

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Octreotide LAR Depot
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less